CLINICAL TRIAL: NCT00282204
Title: Hypnosis Antenatal Training for Childbirth (HATCh): a Randomised Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Women's and Children's Hospital, Australia (Other Government)
Responsible Party: Dr A.M.Cyna, CYWHS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ACTRN012605000018617
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2010-12

CONDITIONS: Pregnancy; Labor
Keywords: Hypnosis; Hypnotherapy; Childbirth; Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Usual care control
- Hypnosis + CD (Experimental): Hypnosis plus audio cd on hypnosis
  Interventions: Behavioral: antenatal hypnosis + audio compact disc on hypnosis
- Audio CD on Hypnosis (Active Comparator): Audio CD on hypnosis sessions weekly on three occasions after 34 weeks gestation
  Interventions: Behavioral: Audio compact disc on hypnosis

INTERVENTIONS:
Behavioral: antenatal hypnosis + audio compact disc on hypnosis
  Arms: Hypnosis + CD
Behavioral: Audio compact disc on hypnosis
  Arms: Audio CD on Hypnosis

SUMMARY:
Antenatal hypnosis is associated with a reduced need for pharmacological interventions during childbirth. This trial seeks to determine the efficacy or otherwise of antenatal group hypnosis preparation for childbirth in late pregnancy.

DETAILED DESCRIPTION:
Background: Although medical interventions play an important role in preserving lives and maternal comfort they have become increasingly routine in normal childbirth. This may increase the risk of associated complications and a less satisfactory birth experience. Antenatal hypnosis is associated with a reduced need for pharmacological interventions during childbirth. This trial seeks to determine the efficacy or otherwise of antenatal group hypnosis preparation for childbirth in late pregnancy.

Methods / Design: A single centre, randomised controlled trial using a 3 arm parallel group design in the largest tertiary maternity unit in South Australia. Group 1 participants receive antenatal hypnosis training in preparation for childbirth administered by a qualified hypnotherapist with the use of an audio compact disc on hypnosis for re-enforcement; Group 2 consists of antenatal hypnosis training in preparation for childbirth using an audio compact disc on hypnosis administered by a nurse with no training in hypnotherapy; Group 3 participants continue with their usual preparation for childbirth with no additional intervention. Women > 34 < 39 weeks gestation, with a singleton, viable fetus, vertex presentation, who are not in active labour or planning a vaginal birth are eligible to participate. Allocation concealment is achieved using telephone randomisation. Participants assigned to hypnosis groups are trained as near as possible to 37 weeks gestation. Group allocations are concealed from treating obstetricians, anaesthetists, midwives and those personnel collecting and analysing data. Our sample size of 135 women / group gives the study 80% power to detect a clinically relevant fall of 20% in the number of women requiring pharmacological analgesia - the primary endpoint. We estimate that approximately 5-10% of women will deliver prior to receiving their allocated intervention. We plan to recruit 150 women / group and perform interim analyses when 150 and 300 participants have been recruited. All participants will be analysed according to the "Intention to treat" principle with comprehensive pre-planned cost- benefit and subgroup analyses.

Discussion: If effective, hypnosis would be a simple, inexpensive way to improve the childbirth experience, reduce complications associated with pharmacological interventions, yield cost savings in maternity care, and provide evidence to guide clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* women > 34 < 39 weeks gestation; singleton, viable fetus, vertex presentation, who are not in active labour (active labour is defined as cervical effacement and dilatation associated with regular uterine contractions) and who are planning a vaginal birth.

Exclusion Criteria:

* Previous hypnosis preparation for childbirth;
* poor understanding of English requiring translator;
* women who are already enrolled in another pregnancy trial where analgesia requirements are an outcome measure;
* active psychological or psychiatric problems such as: active depression requiring treatment by a psychiatrist;
* schizophrenia;
* prior psychosis;
* severe intellectual disability.
* Women with pain caused by specific pathological entities such as: congenital neuromuscular disorders; spina bifida; metastatic disease; osteoporosis; rheumatoid arthritis; fractures,are also excluded

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2005-12; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The use of pharmacological analgesia during labour and childbirth will be collected from the birth register where all analgesia is documented by the attending midwife | Within 24 hours of the birth

SECONDARY OUTCOMES:
1. Maternal rating of the overall pain experienced during labour and childbirth | Usually within 48 hours or before discharge from hospital
2. Mode of delivery | Within 24 hours of the birth
3. Use of oxytocics | Within 24 hours of the birth
4. Postnatal depression | At 6 weeks and 6 months postnatal
5. Maternal anxiety | At 6 weeks and 6 months postnatal
6. Neonatal Apgar score at 5 minutes < 7 | within 24 hours of birth
7. Maternal admission to the High Dependency Unit (HDU) or the Intensive Care Unit (ICU) | within 24 hours of birth
8. Maternal rating whether the birth experience was. Worse / better / same as expected | within 24 hours of birth
9. Maternal rating of control during the labour during the birth | within 24 hours of birth
10. Maternal rating whether the birth was rated positive or negative experience | within 24 hours of birth
11. Length of neonatal nursery stay | within 24 hours of birth
12. Length of maternal stay in hospital | within 6 months of the birth
13. Number of women breast feeding at discharge from hospital and at 6 weeks and 6 months | 6 months after birth

CONTACTS AND LOCATIONS:
Overall Officials: Marion I Andrew, FANZCA, Principal Investigator — Women's and Children's Hospital, Australia; Allan M Cyna, FRCA, Study Director — Women's and Children's Hospital, Australia
Locations (1):
- Women's and Children's Hospital, Adelaide, South Australia, Australia

REFERENCES:
- [Background] Cyna AM, Andrew MI, Robinson JS, Crowther CA, Baghurst P, Turnbull D, Wicks G, Whittle C. Hypnosis Antenatal Training for Childbirth (HATCh): a randomised controlled trial [NCT00282204]. BMC Pregnancy Childbirth. 2006 Mar 5;6:5. doi: 10.1186/1471-2393-6-5. PMID 16515709